CLINICAL TRIAL: NCT05454150
Title: Balloon-Expandable Versus Self-expanding Transcatheter Heart Valve for Treatment of Symptomatic Native Aortic Valve Stenosis
Brief Title: Balloon-Expandable Versus Self-expanding Transcatheter Heart Valve for Treatment of Symptomatic Native Aortic Valve Stenosis (BEST)
Acronym: BEST
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Collaborators: Ministry of Health, France (Other Government); Institut universitaire de cardiologie et de pneumologie de Québec, University Laval (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021_0513; 2021-A02554-37 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2022-07-07; First posted 2022-07-12 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Aortic Valve Stenosis
Keywords: Aortic valve stenosis; TAVI; Balloon-expandable transcatheter heart valve; Self-expanding transcatheter heart valve,; heart valve disease
MeSH Terms: conditions — Aortic Valve Stenosis; Heart Valve Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- TAVI with balloon-expandable valve (Sapien 3/Ultra, Edwards Lifesciences©) (Experimental)
  Interventions: Device: balloon-expandable valve
- TAVI with self-expanding valve (Evolut R/Pro, Medtronic©) (Active Comparator)
  Interventions: Device: self-expanding valve

INTERVENTIONS:
Device: balloon-expandable valve — Sapien 3/Ultra, Edwards Lifesciences©
  Arms: TAVI with balloon-expandable valve (Sapien 3/Ultra, Edwards Lifesciences©)
Device: self-expanding valve — Evolut R/Pro, Medtronic©
  Arms: TAVI with self-expanding valve (Evolut R/Pro, Medtronic©)

SUMMARY:
Over the last years, several randomized studies comparing transcatheter aortic valve implantation (TAVI) to surgical aortic valve replacement (SAVR) have established TAVI as a treatment option in symptomatic patients with aortic stenosis (AS) (1,2,3). Most transcatheter heart valves (THV) available are designed on either a balloon-expandable (BE) or a self-expanding (SE) concept.

Despite major differences, both designs are recommended to be used indifferently in most of the clinical situations and a significant number of centers only implant one of this two THV design. It remains unclear however, whether these 2 very different THV concepts are achieving similar or different clinical outcomes and could be considered a single "Class" of device. While there is an urgent clinical need to clarify this issue in an exponentially growing therapeutic field, to date no large randomized study powered to compare the 2 THV designs on individual endpoints has been conducted or initiated. Recently, two large-scale French registry-based propensity matched analyses, including more than 30,000 patients, have reported a higher 90 days and 1-year mortality with the use of SE as compared to BE-valve (4,5). However, as the propensity-score matching-approach cannot rule out residual confounders, and as some of the most recent THV iterations were not part of the investigation, there is an urgent need to conduct a randomized trial sufficiently powered to compare head-to-head the latest generation of SE and BE-valve on all-cause mortality. In addition, two small randomized studies have recently showed the inferiority of a new SE-valve compared to BE-valve and SE-THV (SCOPE1 trial, J Lanz. Lancet. 2019 Nov 2;394(10209):1619-1628. and SCOPE 2 trial, Circulation in press), thus further questioning wether THV should be considered as a single "Class" regardless the THV design.

The objective of the present randomized clinical investigation will be to evaluate the impact of THV design (SE vs BE) on the risk of all-cause mortality at 90 days and 1 year.

The present clinical investigation will the first randomized clinical investigation to compare head to head the benefit of BE-valve over SE-valve on total mortality and /or disabling stroke at 90 days and 1-year using a superiority design. Previous head-to-head studies included only a small number of patients, non-inferiority designs and combined endpoints. This clinical investigation will be the first to generate sufficient evidences to change clinical practice and international guidelines to clarify whether one THV design is superior (or not) to the other one (BE vs SE-valve). The result of the clinical investigation is key for clinicians indicating the treatment and for the patients receiving the treatment

ELIGIBILITY:
The study population will be comprised of all patients with severe, calcific, symptomatic aortic stenosis eligible to percutaneous transfemoral TAVI with BE or SE-valve according to the investigating center heart team.

The inclusion/exclusion criteria are limited and primarily intend to select patient eligible to both BE and SE-valve. This allows for a study cohort whose composition is expected to be close to an all-comers cohort and therefore representative for the standard TAVI population seen in daily practice.

Inclusion Criteria:

* Symptomatic severe aortic stenosis defined according to the current echocardiography criteria of the European Society of Cardiology guidelines2.
* Heart team of the investigating center agrees that the patient is eligible to TAVI with BE-valve SAPIEN 3 (Edwards Lifesciences©) (or further iterations of the same family) OR TAVI with the SE-valve Evolut-R/pro (Medtronic©) (or futher iterations of the same family).
* Heart team of the investigating center agrees that TAVI is feasible via percutaneous transfemoral approach.
* Written informed consent to the BEST study
* Written informed consent to the FRANCE-TAVI registy
* All valve anatomy are authorized (bicuspid or tricuspid aortic valve)

Exclusion Criteria:

* Age < 18 years old
* Patient with legal protection
* Non-affiliation to a social security scheme
* Pregnancy
* Subject participating in another research protocol on TAVI procedure
* Patients presenting with an anatomy that is regarded unsuitable for the implantation of one of the two valve types
* TAVI through nontransfemoral approach or surgical cutdown
* Valve-in-valve procedure (TAVI in TAVI or TAVI in surgical aortic bioprosthesis)
* Implantation of Accurate Neo or Accurate Neo2 valve (Boston scientific)
* Severe aortic regurgitation (>3+)
* Refusal to participate to FRANCE-TAVI registry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1960 (Actual)
Dates: Start 2023-04-19 (Actual); Primary Completion 2025-10-29 (Actual); Study Completion 2035-12-29 (Estimated)

PRIMARY OUTCOMES:
composite of: device technical failure at exit from procedure room and/or all-cause mortality and/or disabling stroke | at 90-day after TAVI
  An independent clinical event committee (CEC) will adjudicate clinical events according to the VARC-3 definitions.

SECONDARY OUTCOMES:
Composite of device failure, and/or all-cause mortality and/or disabling stroke | at 1 year after TAVI
  An independent clinical event committee (CEC) will adjudicate clinical events according to the VARC-3 definitions.
2Composite of device technical failure, all-cause mortality and/or disabling stroke | At 90 days after TAVI
  An independent clinical event committee (CEC) will adjudicate clinical events according to the VARC-3 definitions.
Device technical failure | at exit from procedure room
  Freedom from mortality, Successful access, delivery of the device and retrieval of the delivery system, Correct positioning of a single prosthetic heart valve into the proper anatomical location, Freedom from surgery or intervention related to the device or to a major vascular or access-related, or cardiac structural complication
Safety | at 90 days after TAVI
  * Technical success at exit from procedure room (VARC 3)*
  * Freedom from all-cause mortality
  * Freedom from all stroke
  * Freedom from VARC type 2-4 bleeding
  * Freedom from major vascular access-related complication
  * Freedom from cardiac structural complication
  * Freedom from acute kidney injury stage 3 or 4
  * Freedom from moderate or severe aortic regurgitation
  * Freedom from new permanent pacemaker due to procedure-related conduction abnormalities
  * Freedom from surgery or intervention related to the device
Device Success | at 90 days after TAVI
  * Technical success at exit from procedure room
  * Freedom from mortality
  * Freedom form surgery or intervention related to the device or to a major vascular or access-related or major cardiac structural complication
  * Intended performance of the valve (mean gradient < 20mmHg, peak velocity <3m/s, Doppler Velocity index ≥ 0.25, and less than moderate aortic regurgitation
Clinical efficacy Clinical efficacy | at 1 year after TAVI
  Ao Technical success at exit from procedure room (VARC 3)*
  * Freedom from all-cause mortality
  * Freedom from all stroke
  * Freedom from hospitalization for procedure- or valve-related causes
  * Freedom from KCCQ Overall Summary Score <45 or decline from baseline of >10 point (i.e. Unfavourable Outcome)
Valve-related clinical efficacy | at 1 year after TAVI
  * Technical success of the TAVI procedure*
  * Intended performance of the valve
  * Freedom from severe PPM at discharge (or 90 days)†
  * Freedom from endocarditis†
  * Freedom from bioprosthesis Valve Failure (BVF)
  * Freedom from stroke or peripheral embolism (presumably valve-related, after ruling out other non-valve aetiologies)
  * Freedom from VARC Type 2-4 bleeding secondary to or exacerbated by antiplatelet or anticoagulant agents, used specifically for valve-related concerns
composite outcome from a patient perspective | AT 90 days and 1 year afet TAVU
  The rate of favourable outcome risk of death
Valve Durability defined as all-cause BVF tricuspid aortic valve | At 90days and 1 year after TAVI
  An independant corelaboratory will review all images. An independent clinical event committee (CEC) will adjudicate clinical events according to the VARC-3 definitions.
11) Stage 2 or 3 hemodynamic valve deterioration | At 1 year after TAVI
  according to VARC-3 n independent clinical event committee (CEC) adjudicate clinical events
device technical failure at exit from procedure room and/or all-cause mortality and/or disabling strok | at 3, 5, 7 and 10 years after TAVI
  according to VARC-3 n independent clinical event committee (CEC) adjudicate clinical events

OTHER OUTCOMES:
1) Rate of patients included in BEST Study successfully matched with the SNDS via the probabilistic linking algorithm of the FRANCE-TAVI registry. | at 1 year after TAVI
  o A successful matching will be defined as >98% of patients of the BEST study successfully matched with SNDS
1) The rate of Hypoattenuated Leaflet Thrombosis (HALT) of any severity as assessed by CT-Scan and transthoracic echocardiography | at 1 year after TAVI
  An independant corelaboratory will review all images

CONTACTS AND LOCATIONS:
Overall Officials: Eric Van Belle, MD,PhD, Principal Investigator — University Hospital, Lille
Locations (21):
- France (21):
  - CH Annecy Genevois, Annecy
  - CHU de Besançon, Besançon
  - CHU de Caen, Caen
  - Hôpital Privé Saint-Martin, Caen
  - CHU de Clermont-Ferrand, Clermont-Ferrand
  - AP-HP Hôpitaux Universitaires Henri Mondor, Créteil
  - CHU de Grenoble, Grenoble
  - Institut Cardiovasculaire Paris Sud, Massy
  - CHU de Montpellier, Montpellier
  - CHU de Nîmes, Nîmes
  - AP-HP Hôpitaux Universitaires Pitié Salpêtrière, Paris
  - Institut Mutualiste Montsouris, Paris
  - CHU de Bordeaux Hôpital Pellegrin, Pessac
  - CHU Reims - Hôpitam Robert Debré, Reims
  - CHU de Saint-Etienne, Saint-Etienne
  - CHU de Nantes - Hôpital Laennec, Saint-Herblain
  - Centre Médico Chirurgical Arnault Tzanck, Saint-Laurent-du-Var
  - CHU de Strasbourg, Strasbourg
  - CHU de Toulouse, Toulouse
  - CHU de Tours, Tours
  - Médipôle Lyon Villeurbanne, Villeurbanne

IPD SHARING:
Plan to Share IPD: No